CLINICAL TRIAL: NCT04949919
Title: Association Between Physical Fitness/Training and Pro-inflammatory/Anti-inflammatory Immune Responses in Patients With End-stage Renal Disease
Brief Title: Physical Fitness/Training and Inflammatory Immune Responses in Patients With End-stage Renal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202000666B0
Record Dates: First submitted 2021-06-07; First posted 2021-07-02 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-05

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESRD patients with supervised training (Experimental): The participants will receive in-hospital supervised exercise training prior to HD
  Interventions: Other: aerobic training by a cycle ergometer and Biodex system 4 pro

INTERVENTIONS:
Other: aerobic training by a cycle ergometer and Biodex system 4 pro — cyclic aerobic training in moderate-intensity and high-intensity interval training plus isokinetic resistance training prior to HD. 60 training sessions in 6 months.

SUMMARY:
The end-stage renal disease (ESRD) leading two causes of death are cardiovascular diseases and sepsis. Exercise improves low physical fitness, available research concerning its effect on the pro-/anti-inflammatory immune response is scarce. In the current proposal, physical fitness is classified into cardiopulmonary fitness and muscle fitness. Muscle fitness is further divided into three domains: strength, mass, and oxidative capacity. The 3-year proposal plan to recruit 90 patients with ESRD who receive regular HD for more than 6 months. Every participant will go through 3 phases：control phase、training phase and the maintenance phase (within-subject design). The hypothesis of the proposal is as follows. (I) When cardiopulmonary fitness/muscle fitness drops to a certain level, the inflammatory immune response will rise. The proposal aims to find the best biomarkers and their cut-off points among the various indicators of cardiopulmonary and muscle fitness that reflect immune dysregulation. (II) Other than physical fitness, cyclic aerobic and resistance training improves pro-/anti-inflammatory immune dysregulation. Additionally, three months after cessation of training, a thorough assessment will be performed to examine whether a healthy lifestyle behavior modification has been achieved and whether the beneficial effect of physical fitness and immune regulation induced by the training program is maintained. The goal of each year is as follows. FIRST year: To explore the relationship between cardiopulmonary fitness and pro-/anti-inflammatory immune response in ESRD patients under HD; SECOND year: To explore the relationship between muscle fitness and pro-/anti-inflammatory immune response; THIRD year: To evaluate the effects of cyclic aerobic and resistance training on physical fitness and pro-/anti-inflammatory immunomodulation in ESRD patients under HD.

DETAILED DESCRIPTION:
In Taiwan, there are more than 90 thousand patients with end-stage renal disease (ESRD) receiving hemodialysis (HD) island-wide. The leading two causes of death are cardiovascular diseases and sepsis. Though evidence is clear that exercise training in this population is beneficial to fitness、quality of life、morbidity, it is seriously underuse. Poor physical fitness is known to associate with high-leveled systemic inflammation and immune dysregulation but the detailed relationship remains unclear in the ESRD population. Moreover, though exercise improves low physical fitness, available research concerning its effect on the pro-/anti-inflammatory immune response is scarce. In the current proposal, physical fitness is classified into cardiopulmonary fitness and muscle fitness. Muscle fitness is further divided into three domains: strength, mass, and oxidative capacity. The 3-year proposal plan to recruit 90 patients with ESRD who receive regular HD for more than 6 months. Every participant will go through 3 phases：control phase、training phase and the maintenance phase (within-subject design). In the control phase, no exercise education or training will be given to the participants. In the training phase, the participants will receive in-hospital supervised exercise training prior to HD. The training program will last 6 months and about 60 training sessions in total. The training protocol contains cyclic aerobic training in moderate-intensity and high-intensity interval training plus isokinetic resistance training. In the following maintenance phase, home-based exercise training will be educated. The control and maintenance phases are 1-2 and 3 months respectively in duration. Before and after each phase and in the middle of the training phase (5-time points totally), every participant will receive a thorough evaluation as follows: CPET with noninvasive cardiac output monitor, isokinetic strength testing, handgrip strength, muscle oxidative capacity, body composition by dual-energy x-ray absorptiometry, Chinese Kidney Disease and Quality of Life questionnaire and international physical activity questionnaire and blood sampling for pro-/anti-inflammatory markers, including chemokine, cytokine, immune cells, and immuno-regulatory microRNAs, etc. The hypothesis of the proposal is as follows. (I) When cardiopulmonary fitness/muscle fitness drops to a certain level, the inflammatory immune response will rise. The proposal aims to find the best biomarkers and their cut-off points among the various indicators of cardiopulmonary and muscle fitness that reflect immune dysregulation. (II) Other than physical fitness, cyclic aerobic and resistance training improves pro-/anti-inflammatory immune dysregulation. Additionally, three months after cessation of training, a thorough assessment will be performed to examine whether a healthy lifestyle behavior modification has been achieved and whether the beneficial effect of physical fitness and immune regulation induced by the training program is maintained. The goal of each year is as follows. FIRST year: To explore the relationship between cardiopulmonary fitness and pro-/anti-inflammatory immune response in ESRD patients under HD; SECOND year: To explore the relationship between muscle fitness and pro-/anti-inflammatory immune response; THIRD year: To evaluate the effects of cyclic aerobic and resistance training on physical fitness and pro-/anti-inflammatory immunomodulation in ESRD patients under HD.

ELIGIBILITY:
Inclusion Criteria:

* on HD for longer than 6 months
* under the permission of their nephrologist
* adequately dialyzed (most recent Kt/V > 1.2) and stable during dialysis in the past 3 months

Exclusion Criteria:

* occurrence of hyperkalemia in the past 3 months
* comorbid medical, physical, and mental conditions that contraindicate exercise
* unstable cardiac conditions (eg, unstable angina, heart failure or symptomatic severe aortic stenosis, etc.)
* disabling orthopedic and neuromuscular diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the association between fitness and immune responses in ESRD patients by cardiopulmonary exercise test | three years
  cardiopulmonary exercise test

SECONDARY OUTCOMES:
To examine the levels of inflammatory chemokines in the circulation of patients by Luminex assay | three years
  Luminex assay

OTHER OUTCOMES:
To detect the levels of anti-inflammatory microRNAs in the circulation of patients by qPCR and pro-/anti-inflammatory immunomodulation | three years
  qPCR assay training and pro-inflammatory/anti-inflammatory immune responses in ESRD patients under HD (longitudinal design

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chun Huang, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan